CLINICAL TRIAL: NCT03248986
Title: Effectiveness of Dry Needling in Improving the Functionality of the Affected Arm in the Patient With Stroke
Brief Title: Dry Needling in Stroke to Improve the Upper Limb Functionality
Status: Completed | Type: Observational
Sponsor: Guadarrama Hospital (Other)
Collaborators: University of San Jorge (Unknown)
Responsible Party: Principal Investigator, J. Nicolas Cuenca Zaldivar, Rehabilitation Service Principal Investigator, Guadarrama Hospital
Other Study IDs: 1.0
Record Dates: First submitted 2017-08-08; First posted 2017-08-15 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Spasticity, Muscle; Functionality; Quality of Life
MeSH Terms: conditions — Muscle Spasticity | interventions — Dry Needling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Dry needling — Dry needling of the spastic muscles of the affected arm through DNHS®.

SUMMARY:
A single-center, observational, prospective, single dynamic cohort study with before-after design. Treatment with 6 sessions using dry needling with DNHS® (Dry Needling for Hypertonicity and Spasticity) on the spastic muscles of the affected arm in patients with stroke. Spasticity will be assessed by Modifying Modified Ashworth Scale (MMAS), functionality with the Fugl-Meyer scale for the upper limb, motor recovery with Brunnstrom Stages Scale (BSS) and upper limb spasticity pattern (ULP), pain by 10-points Numerical Rating Scale (NRS10) and the quality of life with the Euro QoL 5D survey.

DETAILED DESCRIPTION:
Once each patient has signed the informed consent document and it has been verified that the inclusion criteria are met, it will be assigned the same identification number (ID) that is related to its Clinical History (CH) by simple coding; custody of the file with the relationship of each ID with its CH will be the responsibility of the principal investigator.

Patients admitted to the Guadarrama Hospital with the diagnosis of stroke and who meet the eligibility criteria will be treated by their usual physiotherapist, who will administer the standard dry needling intervention.

Patients will receive 6 sessions of DNHS® technique with an interval of 1 week between each session (1st to 4th sessions) and every 15 days (5th and 6th sessions). The procedure will be applied according to the corresponding protocols established in the NWPs (Normalized Work Plans) used in the usual clinical practice in the Guadarrama Hospital.

The DNHS® technique is specifically indicated for the treatment of spasticity. This technique differs from that usually used to relieve pain and deactivate myofascial trigger points (MTPs). The muscles to be treated are placed in a submaximum stretching position; the evaluation criteria when defining the needle insertion zone are based on finding an increase in modularity and muscle activity in the area when the muscle undergoes rapid stretching. Once the area to be treated is located, the needle is inserted and moves between 0.5 and 1 cm in / deep and fan out / surface to cause a local or global spasm reaction. Treatment ceases when the frequency of these responses decreases markedly or disappears. If the patient feels "not tolerable" pain (some discomfort from the dry needling is usual), you can stop the treatment at any time.

Before and after each dry needling session patients will be evaluated by their usual physiotherapist, using the upper limb block of the Fugl-Meyer scale that assesses motor skills and sensitivity of the affected arm, evaluation of pain through NRS10 and assessment of spasticity of muscles to be treated by MMAS. Also, at the beginning, in the 4th session and at the end of the study, the Euro-QoL 5D-5L quality of life survey will be administered, with a license for use. In adition BSS and ULP will be evaluated at the begining and at the end of the study. In each dry needling session, the caliber of the needle used, the number of fast-in and fast-out of the needle and the number of the spasm reactions caused for the purpose of establishing the dose pattern shall be recorded for each treated muscle.

ELIGIBILITY:
Inclusion Criteria:

* They must voluntarily understand and sign the relevant informed consent documents and information sheet, before any evaluation / procedure related to the study is conducted.
* Male or female, ≥ 18 years old at the time of consent.
* Have the diagnosis of hemispheric ischemic or hemorrhagic stroke without excluding other causes (surgical, traumatic, etc ...).
* Show spasticity in the affected upper limb, with an MMAS score of 1-3 in one of the following muscle groups: finger flexors, wrist flexors, elbow flexors, forearm pronators, adductors, or internal rotators of the shoulder.

Exclusion Criteria:

* Presence of stiffness (score of 4 in MMAS) or hypotonia (MMAS of 0).
* Severe cognitive impairment, severe language problems, severe vision or hearing impairments that prevent compression and active patient collaboration during evaluation tests.
* Have received treatment by injection of TBA in the 2 months prior to the start of the study.
* Any medical condition that contraindicates dry needling.
* Present some contraindication for the application of dry puncture: Pregnancy, insurmountable fear of needles, allergy to metals (nickel), presence of lesions in the puncture area, scars, tattoos...

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the diagnosis of stroke entering for the first time at the Hospital Guadarrama
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Upper Limb Scale. | 8 weeks
  Evaluation of the functionality of the affected arm

SECONDARY OUTCOMES:
Modification of Modified Ashworth Scale | 8 weeks
  Assessment of spasticity
Euro QoL 5D quality of life scale | 8 weeks
  Quiality of life evaluation

OTHER OUTCOMES:
Numerical Rating Scale 10-points scale | 8 weeks
  Pain evaluation
Brunnstrom Recovery Stages | 8 weeks
  Upper limb motor recovery.
Upper limb pattern | 8 weeks
  Upper limb spastic pattern.

CONTACTS AND LOCATIONS:
Overall Officials: J. Nicolas Cuenca Zaldivar, Principal Investigator — Guadarrama Hospital
Locations (1):
- J.Nicolas Cuenca Zaldivar, Guadarrama, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No